CLINICAL TRIAL: NCT00087815
Title: Complimentary Hyperbaric Oxygen for Brain Radionecrosis
Brief Title: Hyperbaric Oxygen Therapy in Treating Patients With Radiation Necrosis of the Brain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Barrett Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Supportive Care
Other Study IDs: CDR0000510427; UCMC-02101007
Record Dates: First submitted 2004-07-14; First posted 2004-07-16 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-07

CONDITIONS: Brain and Central Nervous System Tumors; Cognitive/Functional Effects; Radiation Toxicity
Keywords: cognitive/functional effects; radiation toxicity; adult brain tumor; childhood brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Radiation Injuries; Brain Neoplasms | interventions — Dexamethasone; Hyperbaric Oxygenation; Mental Status and Dementia Tests; Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: dexamethasone
Drug: hyperbaric oxygen
Procedure: cognitive assessment
Procedure: magnetic resonance imaging
Procedure: positron emission tomography
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Hyperbaric oxygen may increase blood flow and decrease swelling in areas of the brain damaged by radiation therapy. Giving hyperbaric oxygen therapy together with dexamethasone may be an effective treatment for radiation necrosis of the brain.

PURPOSE: This randomized clinical trial is studying how well hyperbaric oxygen therapy works in treating patients with radiation necrosis of the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

* Obtain pilot data demonstrating the potential for increased benefit when complementing conventional steroid therapy with adjunctive hyperbaric oxygen therapy (HBOT) in patients with brain radionecrosis.
* Estimate the magnitude of benefit of HBOT using objective measures of neurologic function, radiographic imaging, and standardized quality of life measures in these patients.
* Determine, preliminarily, the effect of HBOT on cerebral revascularization using perfusion MRI in these patients.
* Determine the feasibility of performing a large-scale, randomized, controlled study (particularly with regard to patient recruitment and retention) comparing HBOT with conventional steroid therapy.

OUTLINE: This is a pilot, randomized, controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (conventional care only): Patients receive baseline steroid therapy comprising oral dexamethasone 4 times daily. Steroid doses are either increased or decreased per standard protocol during the 90-day treatment period. Patients who demonstrate neurological deterioration at each evaluation (as evidenced by a decrease in Karnofsky performance status score) receive escalating doses of dexamethasone until the maximum daily dose of 32 mg is reached. Patients who reach the maximum daily dose of dexamethasone are removed from the study. Patients also receive anticonvulsant therapy during study therapy.
* Arm II (conventional care and hyperbaric oxygen therapy [HBOT]): Patients receive conventional care as in arm I*. Patients also undergo HBOT once daily, 5 days a week, for 90 days (60 treatments total).

NOTE: *Patients in arm II who reach the maximum daily dose of dexamethasone are not removed from the study.

* Cerebral revascularization study: Five patients from each arm are randomly selected to undergo perfusion MRI before treatment and within 1 week after completion of study therapy to determine the proportion of cerebral neovascularization in each arm.

Patients are evaluated during study by standardized physical examinations, positron emission tomography scans, perfusion MRI, complete neurologic assessment, and standardized, health-related quality of life measures at baseline, at 30-day intervals during treatment, at the end of treatment, and at 1, 2, and 4 months after completion of study therapy.

After completion of study therapy, patients are followed at 1, 2, and 4 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Definitive diagnosis of brain radionecrosis by MRI and positron emission tomography scan

  * Clinically symptomatic with signs of worsening neurologic deficits (e.g., focal deficits or intractable seizures)
* Condition currently managed with increasing steroid dosage

PATIENT CHARACTERISTICS:

* No severe pulmonary disease (i.e., untreated pneumothorax, emphysema, chronic obstructive pulmonary disease, or asthma)
* No active congestive heart failure
* LVEF ≥ 35%
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychological, familial, sociological, or geographical conditions that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior or concurrent bleomycin
* No concurrent doxorubicin hydrochloride
* No concurrent disulfiram

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-09; Study Completion 2005-06

PRIMARY OUTCOMES:
Vasogenic edema volume by MRI at baseline, every 30 days during treatment, at the end of treatment, and then at 1, 2, and 4 months after treatment
Lesion volume (contrast enhancement and necrotic core) by MRI at baseline, every 30 days during treatment, at the end of treatment, and then at 1, 2, and 4 months after treatment
Neurologic status, including mental status, cranial nerves, motor function, sensory function, reflexes, coordination, and gait at baseline, every 30 days during treatment, at the end of treatment, and then at 1, 2, and 4 months after treatment
Health-related quality of life by Short Form-36 Health Survey and General Well-Being Schedule at baseline, every 30 days during treatment, at the end of treatment, and then at 1, 2, and 4 months after treatment
Revascularization by perfusion MRI at baseline, every 30 days during treatment, at the end of treatment, and then at 1, 2, and 4 months after treatment
Survival every 30 days during treatment, at the end of treatment, and then at 1, 2, and 4 months after treatment
Drop-out rate by steroid dosage at baseline, every 30 days during treatment, at the end of treatment, and then at 1, 2, and 4 months after treatment
Tumor progression by physical examination, positron emission tomography scans, and MRI at baseline, every 30 days during treatment, at the end of treatment, and then at 1, 2, and 4 months after treatment
Brain radionecrosis progression by MRI at baseline, every 30 days during treatment, at the end of treatment, and then at 1, 2, and 4 months after treatment
Adverse events (e.g., events related to barotrauma and oxygen or steroid toxicity) at baseline, every 30 days during treatment, at the end of treatment, and then at 1, 2, and 4 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Gesell, MD, Principal Investigator — Barrett Cancer Center
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States